CLINICAL TRIAL: NCT00131183
Title: The Effect of Testosterone Therapy on Angina Threshold and Atheroma in Patients With Chronic Stable Angina
Brief Title: Testosterone Therapy on Angina Threshold and Atheroma in Patients With Chronic Stable Angina
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STH13979
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2006-09

CONDITIONS: Angina Pectoris
Keywords: Angina Pectoris; Arteriosclerosis; Testosterone
MeSH Terms: conditions — Angina Pectoris; Arteriosclerosis | interventions — testosterone undecanoate

INTERVENTIONS:
Drug: Nebido

SUMMARY:
This study aims to address the following questions on the effects of testosterone therapy in men with coronary ischaemia:

* Does the anti-anginal effect persist long term? Many of the published studies are acute single dose trials and none of the chronic studies have assessed patients formally beyond a few months. The investigators' earlier studies were limited to 3 months.
* Does testosterone therapy in men affect the levels of measurable atheroma? There is currently no in-vivo human evidence that androgen therapy inhibits or reduces levels of atheroma, although there is abundant evidence in animals to suggest a potential improvement.

This study addresses the two issues and would be of one-year duration but would be the longest trial of testosterone therapy in men with cardiovascular disease. The primary endpoint is the change in time to ST- segment depression of > 1mm during exercise testing.

DETAILED DESCRIPTION:
In the past 4 years the investigators' research group has completed 2 studies on the effect of testosterone therapy on exercise induced coronary ischaemia (clinically manifest as angina pectoris). We, the investigators at Sheffield Teaching Hospitals, have shown that testosterone replacement therapy improved exercise duration on the treadmill and prolonged time to ischaemia (ischaemic threshold). Moreover, we demonstrated a dose response relationship between the increase in exercise duration and the baseline testosterone level so that men with lower baseline testosterone level derived the greatest symptomatic benefit from replacement therapy. Importantly we have also demonstrated that the effects of testosterone are maintained in the presence of concomitant anti-anginal drug therapy and at physiological levels of testosterone therapy. (English et al. 2000; Malkin 2004)

Furthermore we have found the prevalence of men with coronary disease and low serum testosterone levels to be approximately 25%. This represents a large population of men with low testosterone levels that may benefit symptomatically from testosterone therapy. These men qualify for androgen replacement therapy per se simply to relieve hypogonadal symptoms and maintain bone mineral density and there are clinical guidelines recommending physiological testosterone replacement in this cohort. (Morales and Lunenfeld 2002) The safety issues relating to testosterone treatment which comprise a theoretical increased risk of prostate neoplasia and increased erythropoiesis are of limited relevance in this population because replacement therapy only returns the testosterone level to the physiological range. Indeed, there is no evidence that appropriate testosterone therapy increases the risk of prostate cancer. More importantly, prostate cancer can be identified early by screening for prostate specific antigen allowing careful surveillance during replacement therapy.

This study aims to address the following questions on the effects of testosterone therapy in men with coronary ischaemia:

* Does the anti-anginal effect persist long term? Many of the published studies are acute single dose trials and none of the chronic studies have assessed patients formally beyond a few months. Our earlier studies were limited to 3 months.
* Does testosterone therapy in men affect the levels of measurable atheroma? There is currently no in-vivo human evidence that androgen therapy inhibits or reduces levels of atheroma, although there is abundant evidence in animals to suggest a potential improvement.

This study addresses the two issues and would be of one-year duration but would be the longest trial of testosterone therapy in men with cardiovascular disease.

The primary endpoint is change in time to ST- segment depression of > 1mm during exercise testing.

ELIGIBILITY:
Inclusion Criteria:

* Males over 20 years of age
* Stable, chronic angina pectoris for > 1 month
* ST- segment depression of > 1mm within 12 minutes of the Bruce protocol
* Willing and able to give informed consent and comply with the study protocol
* Serum testosterone (< 12nmol/L)

Exclusion Criteria:

* Use of androgen therapy or anabolic steroids within 6 months of entry into the study (i.e. screening visit/visit 1) or concurrent use of androgens including dehydroepiandrosterone (DHEA), anabolic steroids, clomipramine, antiandrogens, estrogen, cytochrome P450 inducing medicines (e.g. quinidine, ketoconazole, macrolides), corticotrophins (ACTH), oxyphenbutazone
* Contraindication to treatment with Nebido®.
* Organic hypothalamic-pituitary pathology
* Prostate specific antigen (PSA) >= 4ng/ml
* Severe symptomatic benign prostatic hyperplasia
* Patients actively or potentially trying to start a family or requiring fertility treatment
* Suspicion of, current, or past history of breast or prostatic carcinoma
* Myocardial infarction (MI), coronary artery bypass graft surgery (CABG) or percutaneous transluminal coronary angioplasty (PTCA) in the last three months.
* Significant hepatic, respiratory, haematological or renal disease
* Haematocrit > 50% at entry to the study (i.e. screening visit/visit 1)
* History of significant arrhythmia, Wolff-Parkinson-White (WPW) syndrome, > 1st degree heart block, or cerebrovascular accident (CVA) within the last three months
* History of drug or alcohol abuse
* Receiving other trial drugs within 12 weeks
* Hypotension (systolic blood pressure [BP] < 100 mm Hg)
* Severe, malignant, complicated, renovascular, secondary, or uncontrolled hypertension (BP > 180/114)
* Hypercalcaemia
* Nephrotic range proteinuria
* Symptomatic obstructive sleep apnoea syndrome
* Electrocardiogram (ECG) abnormalities that preclude ST- segment analysis (eg left bundle branch block [LBBB], atrial fibrillation [AF])

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in time to ST- segment depression of > 1mm during exercise testing

SECONDARY OUTCOMES:
Change in carotid atheroma assessed by media:intimal thickness ratio of the carotid artery
Change in time to exercise induced chest pain as judged by a single observer
Change in frequency of attacks of angina as recorded in the patients' angina diary
Change in high sensitivity C reactive protein (hs-CRP)
Change in scores on the Seattle Angina Questionnaire (SAQ)
Change in scores of quality of life (Euroquol)
Change in scores of depression using the Beck Depression Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Kevin S Channer, MBChB (Hons), Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom